CLINICAL TRIAL: NCT02427334
Title: Dienogest Versus Luteal Phase Fluoxetine in the Management of Premenstrual Syndrome: A Randomized Double Blind Placebo Controlled Trial
Brief Title: Dienogest Versus Luteal Phase Fluoxetine in the Management of Premenstrual Syndrome
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, AbdelGany Hassan, Lecturer of Gynecology and Obstetrics, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PMS
Record Dates: First submitted 2015-04-20; First posted 2015-04-28 (Estimated); Last update posted 2020-12-01 (Actual); Status verified 2020-11

CONDITIONS: Premenstrual Syndrome
MeSH Terms: conditions — Premenstrual Syndrome | interventions — dienogest; Fluoxetine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Dienogest (Active Comparator): women will receive oral dienogest 2mg for 14 days starting from the 15th day of menstruation
  Interventions: Drug: Dienogest
- Fluoxetine (Active Comparator): women will receive oral fluoxetine 20mg for 14 days starting from the 15th day of menstruation
  Interventions: Drug: Fluoxetine
- Placebo (Placebo Comparator): women will receive oral placebo for 14 days starting from the 15th day of menstruation
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dienogest — women will receive oral dienogest 2mg for 14 days starting from the 15th day of menstruation
  Arms: Dienogest
Drug: Fluoxetine — women will receive oral fluoxetine 20mg for 14 days starting from the 15th day of menstruation
  Arms: Fluoxetine
Drug: Placebo — women will receive oral placebo for 14 days starting from the 15th day of menstruation
  Arms: Placebo

SUMMARY:
Two hundreds and ten women with premenstrual syndrome will be randomly divided into 3 equal groups using computer generated random numbers. Group 1 will receive oral dienogest (visanne® Bayer, Germany) 2mg for 14 days starting from the 15th day of menstruation, Group 2 will receive fluoxetine (Prozac® Lilly, UK) 20mg and group 3 will receive an oral placebo foe 14 days starting from the 15th day of menstruation.

DETAILED DESCRIPTION:
Premenstrual syndrome (PMS) manifests with distressing physical, behavioral and psychological symptoms, in the absence of organic or underlying psychiatric disease, which regularly recur during luteal phase of each menstrual cycle and disappear or significantly improve by the end of menstruation. Approximately 85-90 % of women may experience premenstrual emotional and physical changes in their reproductive age and the prevalence of severe PMS ranges from 3% to 8%.

The etiology of PMS is unknown but cyclical ovarian activity and the effect of estradiol and progesterone on serotonin and gamma-amino butyric acid are key factors. Absence of PMS before puberty, in pregnancy and after the menopause supports a role of cyclical ovarian activity in PMS etiology. PMS symptoms include psychological symptoms like mood swings, irritability, depression and feeling out of control; physical symptoms like breast tenderness, bloating and headaches; and behavioral symptoms like reduced visuospatial and cognitive ability. To diagnose PMS, symptoms should be recorded prospectively over two cycles using a symptom diary. Several symptom diaries exist but the Daily Record of Severity of Problems (DRSP) is reliable and simple for patients.

There is increasing evidence that serotonin may be important in the pathogenesis of PMS. A number of selective serotonin reuptake inhibitors have been used to treat PMS. Fluoxetine at was found to significantly reduce symptoms of tension, irritability and dysphoria, as well as physical symptoms compared with placebo, as measured by visual analogue scales. Luteal phase sertraline was found effective in the management of severe PMS.

Historically, treatment with progesterone was based on the hypothesis that in PMS sufferers, the ratio of progesterone and its derivatives to other hormones was lower than is usual in women. This allowed oestrogens to cause water retention, because there was insufficient progesterone to oppose them.

Gama amino butyric acid (GABA) produced by inhibitory neurons calms symptoms of anxiety, irritability and aggression. Part of the receptors, called GABA(A) on the neurone surface, necessary for GABA to have its effect, cannot be made without the break-down products of progesterone. The occurrence of severe symptoms has been correlated with falling levels of progesterone metabolites. Therefore, progesterone could relieve the symptoms of PMS by preventing falling levels of progesterone metabolites and loss of GABA(A) enhancement.

PMS will be diagnosed prospectively using the DRSP. DRSP is a questionnaire comprised of 25 physical and emotional symptoms including impairment of physical and social activities, women will be asked to give a score of 1 to 6 for each symptom 1 = not at all, 2 = minimal, 3 = mild, 4 = moderate, 5 = severe, 6 = extreme. The investigators will add the symptoms scores of the first day of menses and PMS will be excluded if the score was < 50. If the total score is greater than 50, the patients will record two cycles of symptoms. If more than three items have an average score of more than 3 (mild) during the luteal phase, the investigators will add the scores of five-day intervals during the luteal and follicular phases. PMS will be diagnosed when the luteal phase score is 30 percent greater than the follicular phase score in the 2 months. Women with PMS will be asked to take the drugs for 3 months and keep recording their symptoms and symptom scores will compared to those documented before treatment.

Two hundreds and ten women with premenstrual syndrome will be randomly divided into 3 equal groups using computer generated random numbers. Group 1 will receive oral dienogest (visanne® Bayer, Germany) 2mg for 14 days starting from the 15th day of menstruation, Group 2 will receive fluoxetine (Prozac® Lilly, UK) 20mg and group 3 will receive an oral placebo foe 14 days starting from the 15th day of menstruation.

ELIGIBILITY:
Inclusion Criteria:

* PMS
* Consents to the procedure

Exclusion Criteria:

* Previous medical treatment for PMS
* Body mass index > 35 kg/m2
* Irregular periods
* Medical disorders like diabetes, hypertension, cardiac, liver, kidney or heart disease

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 210 (Estimated)
Dates: Start 2015-04; Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Improvement of DRSP score | Monthly, up to 3 months
  DRSP scores will be documented in each treatment month, the mean score will be compared with the pretreatment score

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo university hospitals, Cairo, Egypt

REFERENCES:
- [Background] Lustyk MK, Widman L, Paschane A, Ecker E. Stress, quality of life and physical activity in women with varying degrees of premenstrual symptomatology. Women Health. 2004;39(3):35-44. doi: 10.1300/J013v39n03_03. PMID 15256354
- [Background] Endicott J, Nee J, Harrison W. Daily Record of Severity of Problems (DRSP): reliability and validity. Arch Womens Ment Health. 2006 Jan;9(1):41-9. doi: 10.1007/s00737-005-0103-y. Epub 2005 Sep 20. PMID 16172836
- [Background] Smith SS, Gong QH, Hsu FC, Markowitz RS, ffrench-Mullen JM, Li X. GABA(A) receptor alpha4 subunit suppression prevents withdrawal properties of an endogenous steroid. Nature. 1998 Apr 30;392(6679):926-30. doi: 10.1038/31948. PMID 9582073